CLINICAL TRIAL: NCT06262412
Title: Clinical Efficacy and Cost-effectiveness of Internet-delivered Cognitive-behaviour Therapy for Children and Adolescents With Body Dysmorphic Disorder: a Randomised Controlled Trial
Brief Title: Internet-delivered Cognitive-behaviour Therapy for Child and Adolescent Body Dysmorphic Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Vastra Gotaland Region (Other Government); Region Skane (Other)
Responsible Party: Principal Investigator, Lorena Fernández de la Cruz, PhD, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-02193-01
Record Dates: First submitted 2024-01-12; First posted 2024-02-16 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Body Dysmorphic Disorders
Keywords: Body dysmorphic disorder; Cognitive-behavior therapy; Exposure and response prevention; Internet
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Intervention Model Description: Multisite parallel-group randomised controlled superiority trial.
Who Masked: Outcomes Assessor
Masking Description: All study personnel who can be blind to study aims/hypotheses and group allocation, will be blind. Assessors conducting post-treatment and follow-up assessments will be external to the research team and blind to study aims/hypotheses and treatment allocation for the full duration of the trial (up to the 6-month follow-up). The assessors will not receive any information about the study design, objectives or treatment conditions in order to maximise the blinding integrity. At each follow-up assessment, participants will be reminded by their assessor to not reveal details about their treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered cognitive-behaviour therapy (ICBT) (Experimental): A therapist-guided, Internet-delivered cognitive-behaviour therapy (ICBT) programme for children and adolescents with BDD.
  Cognitive-behaviour therapy, Exposure and response prevention (ERP)
  Interventions: Behavioral: Internet-delivered cognitive-behaviour therapy (ICBT)
- Internet-delivered relaxation treatment (IRT) (Active Comparator): A therapist-guided, Internet-delivered relaxation treatment (IRT) programme for children and adolescents with BDD.
  Relaxation training (deep breathing, progressive muscle relaxation, imagery)
  Interventions: Behavioral: Internet-delivered relaxation treatment (IRT)

INTERVENTIONS:
Behavioral: Internet-delivered cognitive-behaviour therapy (ICBT) — The intervention is Internet-delivered and therapist-guided, involving both the adolescent and at least one caregiver. It consists of two separate sets of modules, one for the adolescent and one for the caregiver. The intervention consists of 12 modules, delivered over a maximum of 14 weeks.
  The first part includes psychoeducation about BDD and strategies to resolve possible ambivalence towards psychological treatment. The main goal of the treatment is to help the young person to stop avoiding anxiety-provoking situations (e.g., going to school or participating in social situations) by undertaking exposure tasks and to stop doing unhelpful repetitive behaviours and rituals (e.g., excessive mirror-checking, camouflaging), known as response prevention. Every module also contains homework tasks that are meant to be completed between modules and mainly consist of exposure and response prevention (ERP) tasks based on the young person's individual goals.
  Arms: Internet-delivered cognitive-behaviour therapy (ICBT)
Behavioral: Internet-delivered relaxation treatment (IRT) — The intervention is Internet-delivered and therapist-guided, involving both the adolescent and at least one caregiver. It consists of two separate sets of modules, one for the adolescent and one for the caregiver. The intervention consists of 12 modules, delivered over a maximum of 14 weeks.
  The first part includes psychoeducation about BDD, how anxiety and stress are major contributors to BDD symptoms, and that targeting and reducing stress will have a beneficial impact on those symptoms. The main goal of the treatment is to teach the young person to relax in order to cope with anxiety and appearance concerns. The intervention mainly consists of a relaxation treatment and includes different relaxation skills such as deep breathing, progressive muscle relaxation, and imagery (cognitive relaxation). Every module also contains homework tasks that are meant to be completed between modules and mainly consist of relaxation tasks.
  Arms: Internet-delivered relaxation treatment (IRT)

SUMMARY:
The purpose of this trial is to evaluate the clinical efficacy, the cost-effectiveness and the 6-month durability of a therapist-guided, Internet-delivered cognitive-behavior therapy programme for children and adolescents with body dysmorphic disorder.

DETAILED DESCRIPTION:
Primary objective: To determine the clinical efficacy of a therapist-guided, Internet-delivered cognitive-behaviour therapy (ICBT) programme for body dysmorphic disorder (BDD) in reducing BDD symptom severity in children and adolescents with BDD, compared to a control intervention consisting of a therapist-guided, Internet-delivered relaxation treatment (IRT) for BDD.

Secondary objective: To establish the 6-month durability of the treatment effects and to assess the cost-effectiveness of ICBT, compared with IRT, from multiple perspectives and to conduct a health-economic evaluation of ICBT for BDD at the primary endpoint from a health organisation payer, healthcare resource use, and societal perspective.

Type of trial: A multisite parallel-group randomised controlled superiority trial.

Rationale: BDD is a prevalent and impairing disorder that tends to have a chronic course if left untreated. Adolescent-onset BDD is associated with more severe symptoms, greater lifetime comorbidity, and higher rates of attempted suicide compared to adult-onset BDD. Therefore, early intervention is crucial. BDD can be effectively treated with cognitive-behaviour therapy (CBT), although the current evidence is rather weak and more evidence is needed. Furthermore, CBT for BDD is a highly specialised treatment and many young people do not have access to it. ICBT can be a way to increase the availability of an effective, evidence-based treatment for children and adolescents with BDD.

Trial design and methods: Participants will be recruited nationally across Sweden and will be offered 12 modules of therapist-guided ICBT or 12 modules of therapist-guided IRT delivered over 12 weeks. Under certain circumstances, such as illness or holidays, the design allows participants to pause their therapist-support for a maximum of two weeks, which may extend the treatment length to a maximum of 14 weeks. All potential participants will be initially screened via the telephone or at one of the three participating sites. This will be followed by an inclusion/baseline assessment conducted either at one of the three clinics (BUP OCD och relaterade tillstånd, BUP Specialmottagning or BUP Skåne) or, if face-to-face assessments are not feasible, via a secure video application. Participants who are eligible and have consented will be randomised to one of two trial arms. Participants in the comparator group (IRT) will be offered to cross-over to the ICBT intervention after the primary endpoint.

The primary outcome variable: The primary outcome variable is BDD symptom severity measured by the Yale-Brown Obsessive Compulsive Scale modified for BDD, Adolescent version (BDD-YBOCS-A) at the primary endpoint (1-month follow-up post-treatment). Based on BDD-YBOCS-A scores, responder and remission rates at all follow-up points will be calculated. Response will be defined as ≥30% reduction from baseline; full or partial remission will be defined as a score ≤16.

Planned trial sites: The study will be coordinated from the Department of Clinical Neuroscience at Karolinska Institutet (the Sponsor). There will be 3 collaborating study sites: BUP OCD och relaterade tillstånd (Region Stockholm), BUP Specialmottagning (Västra Götalandsregionen), and BUP Skåne (Region Skåne). Each of the three sites will assess and treat participants from their own region, and occasionally from other regions.

Sample: A total of 154 children and adolescents diagnosed with BDD and their primary caregivers.

Statistical methodology and analysis: Data will be analysed using a pre-specified intention-to-treat statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

1. A primary diagnosis of BDD, based on the diagnostic criteria of the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders. Confirmed by the assessor at the inclusion assessment using a semi-structured diagnostic interview. In cases where it is challenging to rule out the presence of actual physical defects that are clearly noticeable (e.g., if the area of concern is the genitalia), we will make a referral to an appropriate service for an expert opinion.
2. A total BDD symptom severity score on the BDD-YBOCS-A ≥24. Confirmed by the assessor at the inclusion assessment.
3. Age between 12 and 17 years. Confirmed by the caregiver/parent and subsequently by the medical record.
4. A minimum of one available caregiver/parent being able to co-participate and support the child/adolescent throughout the treatment. Confirmed by the caregiver/parent at the inclusion assessment.
5. Regular access to a computer connected to the Internet and a mobile phone to receive SMS messages (one of each per family is enough). Confirmed by the caregiver/parent at the inclusion assessment.

Exclusion Criteria:

1. Previous CBT for BDD for a minimum of five sessions with a qualified therapist within the 12 months prior to the inclusion assessment. Confirmed by the caregiver/parent at the telephone screening and/or the inclusion assessment and by the medical record.
2. Simultaneous psychological treatment for BDD or for any psychiatric comorbidity. Confirmed by the caregiver/parent at the telephone screening and/or the inclusion assessment and by the medical record.
3. Initiation, change of dosage or cessation of any selective serotonin reuptake inhibitors (SSRI) or antipsychotic drugs within the six weeks prior to the inclusion assessment. Confirmed by the caregiver/parent at the telephone screening and/or the inclusion assessment and by the medical record.
4. A diagnosis of organic brain disorder, intellectual disability, psychosis, bipolar disorder, eating disorder, severe depression or alcohol/substance dependence. Confirmed by the caregiver/parent at the telephone screening and/or the inclusion assessment, with supplemental information from the semi-structured diagnostic interview and by the medical record.
5. Immediate risk to self or others requiring urgent medical attention or inpatient care, such as suicidality, or repeated self-injurious behaviours. Confirmed by the caregiver/parent at the telephone screening and/or the inclusion assessment.
6. A documented suicide attempt in the last 12 months. Confirmed by the caregiver/parent at the telephone screening and/or the inclusion assessment or by documentation in the medical record.
7. Child/adolescent and caregiver/parent not able to read and communicate in Swedish. Confirmed by the caregiver/parent at the telephone screening and/or the inclusion assessment.
8. Having a close relationship to an already included participant (e.g., sibling, cousin), to avoid being randomised into two different arms, with the risk of information "leaking" between the groups. Confirmed by the caregiver/parent or assessor at the telephone screening and/or at the face-to-face or video conference inclusion assessment.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale Modified for Body Dysmorphic Disorder, Adolescent version (BDD-YBOCS-A) | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  The BDD-YBOCS-A is a clinician-rated, semi-structured interview. It is used to assess BDD symptom severity. It contains twelve items ranging from 0 to 4. It includes five questions on obsessions, five on compulsions, one about insight, and one to measure behavioural avoidance. Range: 0-48, lower scores mean better outcome.

SECONDARY OUTCOMES:
Treatment response and full or partial remission | Post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  Treatment response and full or partial remission rates will be calculated at each follow-up point. Response will be defined as a reduction ≥30% on the BDD-YBOCS-A from baseline. Full or partial remission will be defined as a total score ≤16 on the BDD-YBOCS-A.
Clinical Global Impression - Severity (CGI-S) | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  Used to provide an overall rating of the BDD severity. Clinician-rated. Range: 1-7, lower scores mean better outcome.
Clinical Global Impression - Improvement (CGI-I) | Post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  Used to assess global improvement. Clinician-rated. Range: 1-7, lower scores mean better outcome.
Children's Global Assessment Scale (CGAS) | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  Used to assess global improvement. Clinician-rated. Range: 1-100, higher scores mean better outcome.
Appearance Anxiety Index (AAI) | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  A self-reported measure that covers cognitions and behaviours typical of BDD. Range: 0-40, lower scores mean better outcome.
Short Mood and Feeling Questionnaire - child version and parent version (SMFQ) + additional suicide item (only child/adolescent) | Baseline (week 0), weekly during treatment (week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  Used to assess depressive symptoms and suicidal ideation. Child/adolescent-reported. Range: 0-29, lower scores mean better outcome.
Generalized Anxiety Disorder - 7 item scale (GAD-7) | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  Used to assess anxiety symptoms. Range: 0-21, lower score mean better outcome. Child/adolescent-reported.
Deliberate Self-Harm Inventory - Youth version (DSHI-Y-7) | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  A 7-item self-reported measure to assess the presence and frequency of participants' non-suicidal self-injury. It will help the investigators to assess risk behaviours throughout the trial. Range: 0-7, lower scores mean better outcome.
  At baseline (week 0) the complete DSHI-Y-7 will be administered. At the post-treatment assessment (week 12) and the follow-up assessments, only questions about self-harm during the last month will be asked and not during the last 12 months.
  Range: 0-7, low score means better outcome. Child/adolescent-reported.
CRAFFT (acronym for the key words Car, Relax, Alone, Forget, Friends and Trouble) | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  A short self-reported instrument used to identify substance use and substance use disorder. Range: 0-6, lower scores mean better outcome. Child/adolescent-reported.
Work and Social Adjustment Scale - youth (WSAS-Y) and parent version (WSAS-P) | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  A self-, and parent-reported instrument assessing functional impairment. Range: 0-40, lower scores mean better outcome. Child/adolescent and parent-reported.
Child Health Utility 9D (CHU9D) | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  A self-reported generic preference-based measure of health-related quality of life designed specifically for use in economic evaluation targeting children and adolescents. Range: 9-45, lower score mean better outcome. Child/adolescent-reported.
Trimbos/iMTA Questionnaire for Costs associated with Psychiatric Illness (TiC-P) | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  The TiC-P collects information on healthcare and societal resource use, including for example items on healthcare resource use, medications, school absenteeism, and parental productivity loss. The use of resources will be translated into corresponding costs. No scores as such are available for this measure. Parent-reported.
Working Alliance Inventory - child (WAI-C) and parent version (WAI-P) | After 3 weeks.
  A 6-item scale measuring the child/adolescent and the caregivers/parents perceived working alliance with their therapist. The scale is rated from 1 to 7, yielding a total score of 7-49. Higher scores mean better working alliance. Child/adolescent and parent-reported.
Client Satisfaction Questionnaire (CSQ-8) | Post treatment (week 12).
  Used to assess treatment satisfaction. The scale has 8 items rated from 1 to 4, yielding a total score of 9-36. Higher scores mean more satisfaction. Child/adolescent and parent-reported.
Treatment Credibility and Expectancy Scale (TCES) | After 3 weeks.
  Used to measure treatment credibility or expectancy of treatment outcome. The TCES includes 5 items rated from 0 to 10, yielding a total score of 0-40, where higher scores indicate higher credibility. Child/adolescent and parent-reported.
Patient Exposure/Relaxation Adherence Scale (PEAS/PRAS) | After 4 and 12 weeks.
  The PEAS/PRAS is a 3-item measure of patient adherence to exposure and response prevention (PEAS) or relaxation training (PRAS). The PEAS/PRAS is one single measure but it is adapted to each of the two arms. The PEAS/PRAS has 3 items rated from 0 to 6, yielding a total score of 0-18. Higher scores mean better outcome. For the current trial, the PEAS will be administered as a self-rated version in the ICBT group and the PRAS will be administered as a self-rated version in the control group.
  Child/adolescent-reported.
Treatment preference | Baseline (week 0) and post treatment (week 12).
  Two items will be administered to the caregiver and to the child/adolescent to assess treatment format preference (i.e., if the participant would have preferred to receive Internet-delivered treatment or in-person treatment for his/her symptoms or if it does not matter), as well as how important the participant believe it is to be able to choose which treatment format he/she receives (rated on a 5-point scale). The questionnaire has been developed by the research team.

OTHER OUTCOMES:
Areas of concern and cosmetic procedures | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  Clinicians will ask about areas of concern through a standardized checklist of 28 different parts of the body . They will also ask about current desire for and/or whether the patient had undergone any past cosmetic/surgical procedure related to their BDD concerns. Clinician rated.
School absenteeism | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  Clinicians will ask the participant and the caregiver if the participant has full, partial or no school attendance (i.e., school drop-out) during the last month.
Concurrent interventions | Baseline (week 0), post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  Clinicians will ask the participant questions about medications (type, dose, indication, and time period) and psychological treatment (type, number of sessions, indication, and time period).
BASS platform usage data | Post treatment (week 12).
  Usage data will be extracted from the BASS platform and entered into the trial database. The data includes number of completed modules, number of logins, number of messages sent to the therapist, and the name of the therapist.
Completed modules | Post treatment (week 12).
  In this trial, and for both treatment conditions, the first four modules contain the minimum amount of information required for the participants to understand the treatment rationale and the tasks that they are supposed to carry out. We will report descriptive statistics on the proportion of individuals in each group having completed at least four modules.
Adverse events questionnaire | After 6 weeks, post treatment (week 12), 1-month follow-up, 3-months follow-up, 6-months follow up.
  A questionnaire will be administered to systematically assess adverse events during the trial. The questionnaire is developed by the research team and includes a checklist with expected adverse events based on previous trials as well as a free text box where other, not listed adverse events can be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Fernández de la Cruz, PhD, Principal Investigator — Department of Clinical Neuroscience (CNS), K8, CPF Mataix-Cols,
Locations (3):
- Sweden (3):
  - BUP Specialmottagning, Sahlgrenska Universitetssjukhuset, Gothenburg
  - Barn- och ungdomspsykiatrin, Region Skåne, Malmo
  - BUP OCD och relaterade tillstånd, Stockholm

IPD SHARING:
Plan to Share IPD: No